CLINICAL TRIAL: NCT06792682
Title: Clinical Study to Explore the Safety and Efficacy of Umbilical Cord Blood Mononuclear Cells in Patients With Secondary Poor Graft Function After Hematopoietic Stem Cell Transplantation
Brief Title: The Safety and Efficacy of Umbilical Cord Blood Mononuclear Cells in Patients With Secondary Poor Graft Function After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024098
Record Dates: First submitted 2024-12-27; First posted 2025-01-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Poor Graft Function
Keywords: Secondary poor graft function; Umbilical cord blood mononuclear cells

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical Cord Blood Mononuclear Cells (Experimental)
  Interventions: Biological: Dose escalation; Biological: Dose extension

INTERVENTIONS:
Biological: Dose escalation — Three dose groups are preset. The doses are 2.0×10^6/kg/time, 3.5×10^6/kg/time and 5.0×10^6/kg/ time respectively, in accordance with the "3+3" dose escalation principle, and proceed in turn.
  Each subject receives conventional treatment plus umbilical cord blood mononuclear cells therapy, with 4 consecutive intravenous infusions of umbilical cord blood mononuclear cells at 1 week intervals.
Biological: Dose extension — According to the safety data of dose escalation stage, one dose group is selected for extension.
  Each subject receives conventional treatment plus umbilical cord blood mononuclear cells therapy, with 4 consecutive intravenous infusions of umbilical cord blood mononuclear cells at 1 week intervals.

SUMMARY:
This study is conducted in a prospective, single-center clinical design and is divided into two stages: dose escalation and dose extension. Patients meeting the diagnostic criteria of secondary poor graft function are selected as the study objects. The safety data of umbilical cord blood mononuclear cells in the treatment of secondary poor graft function are obtained through dose escalation stage, and then one dose is selected for dose extension stage to explore the efficacy of umbilical cord blood mononuclear cells in treating secondary poor graft function.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old; gender is not limited.
2. Meet the diagnostic criteria for secondary poor graft function: After 28 days of transplantation, patients who had achieved hematopoietic reestablishment (ANC ≥ 0.5×10^9/L for 3 consecutive days without G-CSF application, PLT ≥ 20×10^9/L for 7 consecutive days without platelet infusion, Hb ≥ 80g/L for 2 consecutive weeks without red blood cell infusion) again developed two or three line cytopenia lasting more than 2 weeks. Bone marrow examination revealed low myelodysplasia, remission of primary disease, complete donor chimeric cells, and no severe graft-versus-host disease (GVHD) or disease recurrence.
3. Eastern Cooperative Oncology Group (ECOG) physical status score ≤ 2 points.
4. Subjects sign informed consent.

Exclusion Criteria:

1. Serious infection not controlled.
2. Active bleeding.
3. Patients with cardiac insufficiency (ejection fraction<50%), or suffering from serious heart disease, including myocardial infarction, cardiac insufficiency, etc.
4. Patients with hepatic and renal insufficiency (total bilirubin>35µmol/L, ALT and AST>2 times of the upper limit of normal; serum creatinine>130µmol/L).
5. Pregnant or lactating women.
6. Concurrent malignant tumors of other organs.
7. Failure to understand or follow the research protocol.
8. Patients participating in other clinical investigations.
9. Other conditions that the investigators consider inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | From date of the last infusion of umbilical cord blood mononuclear cells until the date of end of follow-up, assessed up to 24 months
  Incidence of adverse events

SECONDARY OUTCOMES:
The recovery time of platelet | Two months after the last infusion of umbilical cord blood mononuclear cells
  The first day of 3 consecutive days with PLT ≥ 20×10^9/L without platelet transfusion
The recovery time of neutrophil | Two months after the last infusion of umbilical cord blood mononuclear cells
  The first day of 3 consecutive days with ANC ≥ 0.5×10^9/L without G-CSF application

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, China, Tianjin, Tianjin Municipality, China